CLINICAL TRIAL: NCT07323121
Title: Randomized, Single-blind, Controlled Study of 40 Hz Flickering Stimulation for Insomnia and Other Non-motor Symptoms in Patients With Parkinson's Disease
Brief Title: 40 Hz Flickering for Insomnia in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Collaborators: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-130-K-99-01; 82430045 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-12-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Insomnia
Keywords: Parkinson's disease; insomnia; sleep disorders; 40 Hz flickering; gamma oscillation
MeSH Terms: conditions — Parkinson Disease; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40 Hz flicker light stimulation (Experimental): Parkinson's disease patients with insomnia receiving 40 Hz flicker light stimulation plus standard PD care.
  Interventions: Device: 40 Hz flicker light device
- 100 Hz flicker light stimulation (Sham Comparator): Parkinson's disease patients with insomnia receiving 100 Hz flicker light stimulation plus standard PD care.
  Interventions: Device: 100 Hz flicker light device

INTERVENTIONS:
Device: 40 Hz flicker light device — A visual stimulation device delivering flicker light at 40 Hz. Participants assigned to this intervention receive 30 minutes of 40 Hz flicker light stimulation every night at bedtime for 7 consecutive days, in addition to their stable antiparkinsonian medication. Device parameters, including light intensity and distance, are adjusted according to the protocol to ensure safety and comfort.
  Arms: 40 Hz flicker light stimulation
Device: 100 Hz flicker light device — A visual stimulation device delivering 100 Hz light (e.g., steady or low-frequency light) with similar appearance and intensity as the 40 Hz device. Participants assigned to this intervention receive 30 minutes of control light exposure every night at bedtime for 7 consecutive days, in addition to their stable antiparkinsonian medication.
  Arms: 100 Hz flicker light stimulation

SUMMARY:
This randomized, single-blind, controlled clinical trial aims to evaluate the efficacy and safety of 40 Hz flicker light stimulation for insomnia in patients with Parkinson's disease (PD). Patients with PD and clinically significant insomnia will be randomly assigned in a 1:1 ratio to receive either 40 Hz flicker light or control light for 30 minutes every night at bedtime for 7 consecutive days, in addition to standard antiparkinsonian treatment.

The primary objective is to determine whether 40 Hz flicker light stimulation improves PD-related insomnia as measured by Parkinson's Disease Sleep Scale-2 (PDSS-2). Secondary objectives include evaluating changes in polysomnography-derived sleep parameters, subjective sleep quality, and other non-motor symptoms, as well as assessing the safety and tolerability of the intervention.

This registration specifically covers the Parkinson's disease insomnia cohort of a larger, previously approved multi-cohort protocol that also includes healthy volunteers and primary insomnia patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disorder characterized by both motor and non-motor symptoms. Insomnia and other sleep disturbances are highly prevalent in PD and significantly impair quality of life, yet current pharmacological therapies are often insufficient and may produce adverse effects. There is a clear need for novel, non-pharmacological approaches to improve sleep in PD.

Gamma-band (around 40 Hz) neural oscillations are associated with cortical network activity and may influence sleep regulation, brain adenosine levels, and glymphatic clearance. Flicker light stimulation at 40 Hz has been shown in preclinical and early clinical studies to modulate gamma oscillations and related neurophysiological processes. Based on these findings, 40 Hz visual flicker stimulation may represent a promising, non-invasive strategy for improving insomnia and other non-motor symptoms in PD.

In this single-center, randomized, single-blind, controlled trial, approximately 30 patients with PD and clinically significant insomnia will be enrolled. Eligible participants will be randomly assigned to receive either 40 Hz flicker light stimulation or control light. Participants in the 40 Hz group will receive visual flicker stimulation at 40 Hz for 30 minutes every night at bedtime for 7 consecutive days, using a dedicated light device, in addition to their stable antiparkinsonian medication. Participants in the control group will receive non-40 Hz light of similar intensity and duration under otherwise identical conditions.

Clinical assessments will include PD-specific sleep scales, particularly the Parkinson's Disease Sleep Scale-2 (PDSS-2), general sleep questionnaires such as the Pittsburgh Sleep Quality Index (PSQI), and sleep diaries. Objective sleep parameters, including total sleep time, sleep efficiency, sleep latency, wake after sleep onset, and number of nocturnal awakenings, will be obtained from polysomnography where applicable. Other non-motor symptoms may also be evaluated using standardized scales. Safety assessments will include monitoring of adverse events, vital signs, and visual or ophthalmic discomfort during and after stimulation.

The parent protocol, initially approved in 2022, included healthy volunteers and primary insomnia patients. The present registration focuses exclusively on the Parkinson's disease insomnia cohort introduced by later protocol amendments and does not include the non-PD cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease according to established clinical criteria (e.g., Movement Disorder Society criteria).
* Age between 50 and 75 years.
* Disease duration ≤ 10 years and Hoehn and Yahr stage ≤ 3 in the "on" state.
* Clinically significant insomnia, defined as Parkinson's Disease Sleep Scale-2 (PDSS-2) total score ≥ 18 points and/or meeting diagnostic criteria for insomnia.
* Stable antiparkinsonian medication regimen for at least 4 weeks prior to enrollment.
* Able and willing to comply with study procedures and provide written informed consent.

Exclusion Criteria:

* Secondary insomnia primarily due to severe systemic diseases or major psychiatric disorders (e.g., psychosis, severe depression or anxiety) or substance abuse.
* History of epilepsy, photosensitive seizures, photosensitive dermatitis, or other conditions in which flicker light stimulation is contraindicated.
* Severe visual impairment or eye diseases that would interfere with light stimulation or safety assessment.
* Unstable or severe medical conditions (e.g., uncontrolled cardiovascular, hepatic, renal, or endocrine disease) that, in the investigator's opinion, make participation unsafe.
* Participation in another interventional clinical trial within the past 3 months.
* Inability to complete study procedures or follow-up due to cognitive, physical, or social reasons.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Parkinson's Disease Sleep Scale-2 (PDSS-2) total score (0-60 points; higher scores indicate worse sleep disturbance). | Baseline and Day 7
  The Parkinson's Disease Sleep Scale-2 (PDSS-2) is a 15-item questionnaire assessing nocturnal symptoms in Parkinson's disease. Each item is scored from 0 to 4, yielding a total score from 0 to 60 points. Higher scores indicate more severe sleep disturbance. The outcome measure is the change in PDSS-2 total score from baseline to Day 7 after the intervention, and the between-group difference (40 Hz vs control) in mean change will be compared.

SECONDARY OUTCOMES:
Change in Parkinson's Disease Sleep Scale-2 (PDSS-2) total score at follow-up (0-60 points; higher scores indicate worse sleep disturbance). | Baseline, Day 7, and Day 28
  The Parkinson's Disease Sleep Scale-2 (PDSS-2) total score ranges from 0 to 60 points, with higher scores indicating more severe sleep disturbance. The outcome measure is the change in PDSS-2 total score from baseline to Day 7 and to Day 28, and the between-group differences (40 Hz vs control) in these changes will be analyzed.
Change in Non-Motor Symptoms Scale (NMSS) total score (0-360 points; higher scores indicate more severe non-motor symptoms). | Baseline and Day 7
  The Non-Motor Symptoms Scale (NMSS) is a clinician-rated instrument assessing the severity and frequency of non-motor symptoms in Parkinson's disease. The total score ranges from 0 to 360 points, with higher scores indicating more severe non-motor symptom burden. The outcome measure is the change in NMSS total score from baseline to Day 7 between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Haochen Sun, Principal Investigator — Jiangsu Province Nanjing Brain Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data that underlie the results of this trial (after de-identification) may be shared upon reasonable request to the principal investigator after publication of the main results, subject to ethics committee approval and institutional regulations.